CLINICAL TRIAL: NCT06857097
Title: Single Anastomosis Sleeve Jejunal Bypass Versus One Anastomosis Gastric Bypass in Management of Morbid Obese Patients: A Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ashraf Gamal Abdelraoof, assistant lecturer of general surgery at sohag university hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-25-2-4MD
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Single Anastomosis Sleeve Jejunal Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single anastomosis sleeve jejunal bypass group (Active Comparator)
  Interventions: Procedure: single anastomosis sleeve jejunal bypass
- one anastomosis gastric bypass (Active Comparator): dissection started just distal to the crows' foot till reaching the lesser sac. A long narrow gastric pouch was created by the endostapler. After that, a longitudinal gastrojejunostomy (4-cm wide) was created at 200 cm distal to the Treitz ligament as the SASJ grou p.
  Interventions: Procedure: One anastomosis gastric bypass

INTERVENTIONS:
Procedure: single anastomosis sleeve jejunal bypass — sleeve was created starting devascularization of greater gastric curve 6 cm proximal to pylorus. Devascularization was done via either a harmonic scalpel or a ligasure device. Dissection was continued proximally till reaching the left diaphragmatic crus. Afterwards that the stomach was resected along the greater curvature via an endostapler over a 36-Fr bougie. After creating the sleeve, two meters of the small bowel were counted starting from the ligament of Treitz, and an antecolic isoperistaltic gastrojejunostomy (4-cm wide) was created with the antrum via linear stapler, and the anterior wall defect was closed by sutures.
  Arms: single anastomosis sleeve jejunal bypass group
Procedure: One anastomosis gastric bypass — dissection started just distal to the crows' foot till reaching the lesser sac. A long narrow gastric pouch was created by the endostapler. After that, a longitudinal gastrojejunostomy (4-cm wide) was created at 200 cm distal to the Treitz ligament as the SASJ group.
  Arms: one anastomosis gastric bypass

SUMMARY:
This study was conducted aiming to assess the efficacy of SASJ bypass as a novel bariatric procedure in terms of operative time, weight loss, complications and effect on comorbidities compared to the outcomes of OAGB within two years after operation.

DETAILED DESCRIPTION:
This study is going to be prospectively randomized. There will be one hundred people with morbid obesity undergoing bariatric surgery at the hospitals of Sohag University and Ainshams University. The investigator will select which individuals will have gastric bypass surgery after counseling patients about all bariatric procedures. The patients were randomly assigned to two equal groups (50 per group); the first patient was OAGB (group A), and the second was SASJ (group B). After the study has been approved by the ethics council of the Sohag University and Ain shams university, Faculty of Medicine, all patients must give written informed consent for participation.

the investigators included a total of 100 cases in this prospective randomized study, and they were divided into two equal groups; SASJ and OAGB groups. The two procedures were performed by the same surgical team adapting standardized techniques. Weight loss parameters were our primary objectives, while secondary outcomes included operative time ,post-operative complications, nutritional(macro and micro nutrients) status, improvement/resolution of comorbidities and quality of life.

Total number of 100 patients, aged between 16 and 60 years, with BMI > 40 kg/m2, or BMI > 35 kg/m2 with the presence of obesity related comorbidity (diabetes mellitus, hypertension, OSAS, osteoarthritis) were enrolled in this study.

An informed written consent was signed by all patients, after complete explanation of the idea of the study, along with the benefits and drawbacks of each procedure. Detailed history taking, physical examination, routine preoperative laboratory investigations and abdominal ultrasonography were performed for all cases.

The 100 cases were randomly allocated into two equal groups SASJ and OAGB groups. Randomization was done in the operating room . All cases were performed by laparoscopy under general anesthesia. The two procedures were performed by 5 ports, .

For the SASJ group , sleeve was created starting devascularization of greater gastric curve 6 cm proximal to pylorus. Devascularization was done via either a harmonic scalpel or a ligasure device. Dissection was continued proximally till reaching the left diaphragmatic crus. Afterwards that the stomach was resected along the greater curvature via an endostapler over a 36-Fr bougie. After creating the sleeve, two meters of the small bowel were counted starting from the ligament of Treitz, and an antecolic isoperistaltic gastrojejunostomy (4-cm wide) was created with the antrum via linear stapler, and the anterior wall defect was closed by sutures.

In the OAGB group .dissection started just distal to the crows' foot till reaching the lesser sac. A long narrow gastric pouch was created by the endostapler. After that, a longitudinal gastrojejunostomy (4-cm wide) was created at 200 cm distal to the Treitz ligament as the SASJ group.

For all procedures, intraoperative methylene blue test was done and an abdominal drain was inserted at the gastric staple line. After operation, all cases were transferred to the internal ward, and started oral intake 6 hours after surgery. Most cases were discharged on the 1st or 2nd post operative day after fully mobilized and appropriate oral intake. Patients were recommended to receive a liquid diet for the first week, followed by soft diet for the following three weeks. There after, a long-term solid diet (hypo-caloric, protein-enriched) was recommended. Daily oral supplements of multivitamins and weekly administration of the intramuscular vitamin B12 were commenced for all cases.

Regular follow up was scheduled for all cases for weekly in the first month then 3, 6 , 12 , 24 months after surgery. During these visits, patients were clinically and biochemically assessed. Any post-operative complications were noted and recorded. Weight changes were recorded as the percentage of excess weight loss (%EWL) and percentage of total weight loss (%TWL).

Our primary outcomes were the %EWL and %TWL, while secondary outcomes included post-operative complications, improvement/resolution of comorbidities.. Diabetes resolution was defined according to Buse et al. as the presence of normal glucose and Hba1c levels in the absence of antidiabetic medications [23], whereas resolution of OSAS was defined by STOPBANG questionnaire with score less than 2 after operation [24]. Hypertension improvement was defined as blood pressure < 140/90 with reduction of medication dose and remission without its cessation [25]. De novo GERD was defined as the post-operative development of reflux symptoms in patients not suffering from it [26], and reflux was confirmed by endoscopy in these cases.

ELIGIBILITY:
Inclusion Criteria:

1. body mass index of over 35 plus the comorbidity presence.
2. body mass index of over 40 with/without comorbidity.
3. patients' willingness to participate in the study.
4. patients' cooperation in follow-up researches.
5. lacking any psychiatric disease.

Exclusion Criteria:

1. Patients negating to change their lifestyle.
2. drug abuse and/or addiction.
3. eating disorder background (e.g., bulimia nervosa).
4. Patients with contraindications to laparoscopic surgery and (or) unfit for surgery.
5. pregnant patients.
6. previous upper abdominal procedures,
7. reflux symptoms
8. major unstable psychiatric illness.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss parameters | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: sohag university hospital, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided